CLINICAL TRIAL: NCT00889252
Title: A Single-Center, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study Evaluating the Safety of a Novel Contact Lens Used Daily in Healthy, Normal Volunteers
Brief Title: Safety Study of a Contact Lens With Ketotifen in Healthy, Normal Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-4539
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- K-Lens (Experimental): Ketotifen combination drug-device product: contact lens (device) and anti-allergy drug
  Interventions: Device: contact lens with ketotifen
- Placebo Lens (Placebo Comparator): Placebo lens
  Interventions: Device: contact lens

INTERVENTIONS:
Device: contact lens with ketotifen — K-Lens (generic name not established) and Ketotifen combination drug-device product
  Arms: K-Lens
Device: contact lens — Placebo contact lens
  Arms: Placebo Lens

SUMMARY:
The purpose of this study is to evaluate the safety of a novel contact lens in healthy normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy normal, soft contact lens wearing volunteers
* normal ocular health
* contact lens correction from +6.00 to -12.00D in each eye and astigmatism of -1.00D or less in each eye

Exclusion Criteria:

* active ocular infection
* history of ocular surgery
* use of topical ophthalmic preparations (including rewetting drops)
* pregnancy or lactation

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pall, OD, MS, FAAO, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Lens: contact lens without drug
Period: Overall Study
Arm/Group | K-Lens | Placebo Lens
Started | 168 | 82
Completed | 161 | 78
Not Completed | 7 | 4
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | K-Lens | Placebo Lens | Total
Number analyzed (Participants) | 168 | 82 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (12.48) | 29.3 (10.77) | 31.5 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 46 | 163
  Male | 51 | 36 | 87
Region of Enrollment [Number; unit: participants]
  United States | 168 | 82 | 250

OUTCOME MEASURES:

1. Primary Outcome: Lid and Lid Margin Erythema, Change From Baseline
Description: Assessment of lid redness using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

2. Primary Outcome: Lid and Lid Margin Swelling, Change From Baseline
Description: Assessment of lid swelling using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

3. Primary Outcome: Conjunctival Redness, Change From Baseline
Description: Assessment of conjunctival redness using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | -0.3 (0.67) | -0.1 (0.58)

4. Primary Outcome: Conjunctival Chemosis, Change From Baseline
Description: Assessment of swelling of the conjunctiva using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

5. Primary Outcome: Corneal Edema, Change From Baseline
Description: Assessment of corneal swelling using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

6. Primary Outcome: Corneal Erosion, Change From Baseline
Description: Assessment of corneal erosion using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

7. Primary Outcome: Corneal Endothelial, Change From Baseline
Description: Assessment of the posterior cornea using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

8. Primary Outcome: Lens Pathology, Change From Baseline
Description: Assessment of the clarity of the intraocular lens using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0.23) | 0 (0.20)

9. Primary Outcome: Flare in Anterior Chamber, Change From Baseline
Description: Assessment of visible protein in the anterior chamber using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

10. Primary Outcome: Cells in Anterior Chamber, Change From Baseline
Description: Assessment of visible cells in the anterior chamber using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

11. Primary Outcome: Corneal Staining - Nasal, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the region towards the nose, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0.27) | 0 (0.24)

12. Primary Outcome: Corneal Staining - Temporal, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the region towards the edge of the face, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0.20) | 0 (0.22)

13. Primary Outcome: Corneal Staining - Inferior, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the bottom region, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | -0.1 (0.51) | 0.0 (0.43)

14. Primary Outcome: Corneal Staining - Superior, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the upper region, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0.13) | 0 (0)

15. Primary Outcome: Corneal Staining - Central, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the central region, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0.19) | 0 (0.19)

16. Primary Outcome: Intraocular Pressure - Change From Baseline
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: mm of mercury
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
mm of mercury | 0.8 (2.45) | 0.6 (2.51)

17. Primary Outcome: Dilated Ophthalmoscopy - Fundus, Change From Baseline
Description: Assessment of changes in abnormalities on the back part of the eye, using the scale: 0=none, 0.5=trace, 1=mild, 2=moderate, 3=severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

18. Primary Outcome: Dilated Ophthalmoscopy - Vitreous, Change From Baseline
Description: Assessment of changes in the vitreous (gel-like fulid of the eye), using the scale: 0=none, 0.5=trace, 1=mild, 2=moderate, 3=severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Units on a scale | 0 (0) | 0 (0)

19. Primary Outcome: Visual Acuity Assessment
Description: Visual acuity was assessed by the investigator using a Snellen visual acuity chart. This outcome counts the number of eyes that had vision of 20/40 or better at the 12 week visit.
Time Frame: at the 12 week visit
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | K-Lens | Placebo Lens
Number analyzed (Participants) | 158 | 75
Number analyzed (eyes) | 316 | 150
Eyes | 316 | 150

ADVERSE EVENTS:
Arm/Group | K-Lens | Placebo Lens
Serious Adverse Events (participants affected / at risk) | 1/168 | 0/82
Other Adverse Events (participants affected / at risk) | 12/168 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | K-Lens (N=168) | Placebo Lens (N=82)
Benign adenoma (Reproductive system and breast disorders) | 1 (1) | 0 — Benign tumor on an ovary, unrelated to test article.
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 — Gallstones, unrelated to test article.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-Lens (N=168) | Placebo Lens (N=82)
Instillation Site Irritation (Eye disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish or publicly present the results of the study without the prior written approval of the sponsor.